CLINICAL TRIAL: NCT01488604
Title: Efficacy and Safety of an Antiviral Polymeric Nasal Spray: A Randomized, Parallel Group, Double-blind, Placebo-controlled Study in Subjects With Early Symptoms of Common Cold
Brief Title: A Study of an Experimental Nasal Spray in Subjects With Early Signs of the Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POCEXP0003; CIV-GB-11-12-003243 (Other: MHRA)
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNS (Experimental): 2 sprays of experimental nasal spray per nostril 4 times per day for 7 days
  Interventions: Device: Polymeric Nasal Spray
- SNS (Sham Comparator): 2 sprays of sham nasal spray per nostril 4 times per day for 7 days
  Interventions: Device: Sham Nasal Spray

INTERVENTIONS:
Device: Polymeric Nasal Spray — Experimental nasal spray
  Other Names: Not yet marketed polymeric nasal spray
  Arms: PNS
Device: Sham Nasal Spray — Sham nasal spray
  Other Names: Not marketed sham comparator
  Arms: SNS

SUMMARY:
This study will test 200 people to see if an experimental nasal spray has an effect on symptoms of the common cold if used when the symptoms start. At the first visit to the clinic, potential subjects will have tests to make sure they qualify to participate in the study.

If they qualify, they will have an equal chance of receiving the experimental nasal spray or a sham nasal spray (one that does not have the experimental formula). At the first visit, subjects will receive their assigned nasal spray and use it once at the clinic. They will also receive a booklet called a diary. Subjects will take the rest of their treatments for day 1 at home, and for the next six days, they will use the nasal spray four times per day and record their symptoms in the diary, as instructed. Then subjects will come back to the clinic for a final visit.

DETAILED DESCRIPTION:
This is an investigation in healthy subjects with early signs of common cold. Subjects will be randomly assigned in a 1:1 ratio to receive either Polymeric Nasal Spray or a matching placebo nasal spray.

Subjects will be screened for eligibility and randomized to treatment at the Screening/ Randomization Visit (Day 1). Subjects will apply the first dose of the nasal spray at this visit under supervision. The other applications will take place at home on Day 1. On Days 2 through 7, subjects will use their assigned nasal spray as 2 sprays per nostril, 4 times per day.

One Follow up Visit will be conducted within 3 days of the last application of nasal spray.

Enrollment will continue until 200 subjects have completed the investigation (100 per treatment group). The subject and the investigative staff will be blinded to the assigned nasal spray.

Efficacy will be measured, and recorded in the subject's diary, and safety will be assessed by reported AEs and ADEs.

ELIGIBILITY:
Inclusion Criteria:

* Have early signs of a common cold: If female of child-bearing potential, have a negative pregnancy test at Screening.
* Have signed and dated the informed consent document, indicating that they have been informed of all pertinent aspects of the investigation
* Are willing and able to comply with scheduled visits, treatment plan, and other investigation procedures

Exclusion Criteria:

* Have had common cold or flu-like symptoms outside the protocol-specified parameters.
* Are current smokers as defined by the protocol.
* Have any medical history or condition or use any drug or device that (per protocol or in the opinion of the investigator) might compromise subject safety, participation in the trial, action of the investigational device, or results of the investigation..
* Are related to anyone involved with the conduct of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Symptoms of the Common Cold | Within 7 days
  Subjects will score their symptoms of the common cold including local symptoms (sore throat, blocked nose, runny nose, cough, and sneezing) and systemic symptoms (headache, muscle ache, and chilliness) on a scale of 0-3, where 0=: None (symptoms not present in the previous 24 hours) and 3= Severe (symptoms disturbing/irritating most of the time).

SECONDARY OUTCOMES:
Effect of Common Cold on Daily Activities | Within 7 days
  Subjects will score how their cold affects daily activities on a scale of 0-3, where 0= None (able to carry out daily activities as normal) and 3= Severe (very limited or no ability to carry out daily activities).
Effect of Common Cold Symptoms on Sleep | Within 7 days
  Subjects will score how their cold affects ability to sleep on a scale of 0-3, where 0= None (no effect on sleep) and 3= Severe (sleep severely affected, or sleep not possible).
Number of Days Lost | Within 7 days
  The number of days lost at school or work because of the common cold will be recorded in the subject diary.
Treatment Outcome | Within 7 days
  Treatment outcome will be recorded by the subject on the evenings of treatment days on a scale of 0-4, where 0=Complete recovery and 4=Deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (3):
- United Kingdom (3):
  - Synexus Thames Valley, Reading, Berkshire
  - Synexus Wales, Cardiff, Llaishen
  - Common Cold Center and Healthcare Clinical Trials, Cardiff, Wales